CLINICAL TRIAL: NCT00485264
Title: A Phase I/II, Multicenter, Open-Label, Noncomparative Study of the International Maternal, Pediatric, Adolescent AIDS Clinical Trials (IMPAACT) Group to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Raltegravir (Isentress, MK-0518) in HIV-1 Infected Children and Adolescents
Brief Title: Safety and Pharmacokinetics (PK) of Raltegravir in HIV (Human Immunodeficiency Virus)-Infected Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1066; 10495 (Registry Identifier: DAIDS ES); IMPAACT P1066 (Other: IMPAACT)
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Suspensions

ARMS (6):
- Cohort I (Experimental): Participants between the ages of 12 and 18 years; receiving raltegravir poloxamer film coated tablet:
  Stage I starting dose: Weight based dose of ~6 mg/kg based on protocol dosing table, taken orally twice daily.
  Final Selected Dose: 400-mg tablet taken orally twice daily.
  Interventions: Drug: Raltegravir poloxamer film coated tablet
- Cohort IIA (Experimental): Participants between the ages of 6 and 11 years, receiving raltegravir poloxamer film coated tablet:
  Stage I starting dose: Weight based dose of ~8 mg/kg based on protocol dosing table, taken orally twice daily.
  Final Selected Dose: 400-mg tablet taken orally twice daily for participants weighing at least 25 kg. Participants < 25 kg were switched to a weight-based dose of the chewable tablet.
  Interventions: Drug: Raltegravir poloxamer film coated tablet
- Cohort IIB (Experimental): Participants between the ages of 6 and 11 years; receiving raltegravir chewable tablet:
  Stage I starting dose: Weight based dose of ~8 mg/kg based on protocol dosing table, taken orally twice daily.
  Final Selected Dose: Weight based dose of ~6 mg/kg according to the dosing table, to a maximum dose of 300 mg, taken orally twice daily.
  Interventions: Drug: Raltegravir chewable tablet
- Cohort III (Experimental): Participants between the ages of 2 and 5 years; receiving raltegravir chewable tablet:
  Stage I starting dose: Weight based dose of ~6 mg/kg based on protocol dosing table, taken orally twice daily.
  Final Selected Dose: Weight based dose of ~6 mg/kg according to the dosing table, to a maximum dose of 300 mg, taken orally twice daily.
  Interventions: Drug: Raltegravir chewable tablet
- Cohort IV (Experimental): Participants between the ages of 6 and 23 months; receiving raltegravir oral granules for suspension (20 mg/mL):
  Stage I starting dose: Weight based dose of ~6 mg/kg orally every 12 hours according to dosing table in protocol or the dose determined by review of all available data.
  Interventions: Drug: Raltegravir oral granules for suspension (20 mg/mL)
- Cohort V (Experimental): Participants between the ages of 4 weeks and 5 months; receiving raltegravir oral granules for suspension (20 mg/mL):
  Stage I starting dose: Weight based dose of ~6 mg/kg orally every 12 hours according to dosing table in protocol or the dose determined by review of all available data.
  Interventions: Drug: Raltegravir oral granules for suspension (20 mg/mL)

INTERVENTIONS:
Drug: Raltegravir poloxamer film coated tablet — Final Selected Dose: 400-mg tablet taken orally twice daily.
  Other Names: Isentress
  Arms: Cohort I
Drug: Raltegravir chewable tablet — Final Selected Dose: Weight based dose of ~6 mg/kg according to the dosing table, to a maximum dose of 300 mg, taken orally twice daily.
  Other Names: Isentress
  Arms: Cohort IIB; Cohort III
Drug: Raltegravir oral granules for suspension (20 mg/mL) — Weight based dose of ~6 mg/kg orally every 12 hours according to dosing table in protocol or the dose determined by review of all available data.
  Other Names: Isentress
  Arms: Cohort IV; Cohort V
Drug: Raltegravir poloxamer film coated tablet — Final Selected Dose: 400-mg tablet taken orally twice daily for participants weighing at least 25 kg. Participants < 25 kg were switched to a weight-based dose of the chewable tablet.
  Other Names: Isentress
  Arms: Cohort IIA

SUMMARY:
Integrase is 1 of 3 HIV (Human Immunodeficiency Virus)-1 enzymes required for viral replication. Raltegravir is a drug that prevents integrase from working properly. This drug has been tested for safety and efficacy in adults, but this is the first study to examine raltegravir in children and adolescents. The purpose of this study was to determine the appropriate dose for raltegravir across the pediatric age range from 4 weeks to 18 years of age, by acquiring short and long term safety data, intensive and population pharmacokinetic (PK) data, and efficacy experience with raltegravir in HIV-infected children and adolescents.

DETAILED DESCRIPTION:
Integrase is one of three enzymes necessary for HIV replication. Integrase allows for the integration of HIV DNA (deoxyribonucleic acid) into the human genome. Raltegravir is a strong and selective inhibitor of HIV integrase. In adults, raltegravir has shown significant antiretroviral activity in clinical trials and is well tolerated. The purpose of this study was to determine the appropriate dose for raltegravir across the pediatric age range from 4 weeks (30 days) to 18 years of age, by acquiring short and long term safety data, intensive and population PK data, and efficacy experience with raltegravir in treatment-experienced, HIV-infected children and adolescents.

The study consisted of two sequential Stages: I and II. The dose finding period of Stage I was intended to examine the pharmacokinetics and short term tolerability and safety of raltegravir in a limited number of participants to permit dose selection for further study in Stage II. The dose finding algorithm required a preliminary assessment of data from the first 4 patients of each cohort (termed a "mini-cohort"). Failure to meet PK targets required dose adjustments, contingent upon the mini-cohort's dose having met safety criteria, followed by reassessment of safety and PK data from the new mini-cohort dose. When a mini-cohort dose had passed both safety and PK criteria, further accrual to and an assessment of results from the full cohort could occur. Again, failure to meet PK targets required dose adjustments contingent upon the full cohort's dose having met safety criteria with subsequent PK and safety evaluation of data from a new cohort taking the new dose.

Chronic dosing, which includes Stage I extension (the period after Stage I dose finding) and Stage II (additional participants enrolled), was intended to provide longer term safety and antiviral activity data in a larger sample of participants. Participants accrued into Stage I and treated only at the dose ultimately selected for their cohorts were combined with those accrued into Stage II, where all patients received only the final selected doses for their respective cohorts. This group is denoted as the Final Dose Population, and results from this group are considered primary, since they reflect only the age-specific doses proposed for commercial use. The group with all participants exposed to raltegravir (at any dose) is denoted as the All Treated Population.

Stage I lasted for a minimum of 48 weeks, Stage II was for 48 weeks, and a long-term follow-up period lasted for 5 years from initial exposure (i.e., 48 weeks of treatment plus 4 years of follow-up). Participants were stratified by age and assigned to one of six cohorts. Participants in Cohort I were between the ages of 12 and 18 years and received poloxamer film coated raltegravir tablets. Participants in Cohort IIA were between the ages of 6 and 11 years, weighed at least 25 kg, and received poloxamer film coated raltegravir tablets. Participants in Cohort IIB were between the ages of 6 and 11 years and received chewable raltegravir tablets. Participants in Cohort III were between the ages of 2 and 5 years and received chewable raltegravir tablets. Participants in Cohort IV were between the ages of 6 months (defined as 180 days) and 23 months and received oral granules for suspension. Participants in Cohort V were between the ages of 4 weeks (defined as 30 days) and 5 months and received oral granules for suspension.

Enrollment for Stage I of this study began with Cohort I and progressed to the other cohorts once preliminary dosage had been determined and safety data were reviewed. When this information had been determined for Cohort I, Cohorts IIA and IIB began enrollment. Once safety and dose data for these cohorts were reviewed, enrollment into Cohort III began. Once safety and dose data for Cohort III were reviewed, enrollment into Cohort IV began and once safety and dose data for Cohort IV were reviewed, enrollment into Cohort V began.

During Stage II of this study, participants took raltegravir at the dosage determined as safe and reaching PK targets based on the the Stage I data. The purpose of Stage II was to determine long-term safety of raltegravir once a safe dose meeting PK targets has been determined.

Participants whose Stage I dose was different from the dose determined for Stage II and who had not had individual dose adjustments because of extreme PK values had their raltegravir dose changed to the selected Stage II dose once it was determined. If individualizing the dose for participants in this manner resulted in a dose increase, these participants had an additional safety visit 4 weeks after the dose modification, and then continued on study visits with no further changes in the visit schedule.

There were at least 9 study visits for participants in this study, occurring during the 48-week raltegravir treatment period. For participants who completed 48 weeks of study and appeared to have benefited from receiving study drug, raltegravir was provided until five years after initial raltegravir exposure. For participants who opted to continue on study-provided raltegravir, extended provision of drug was implemented as part of a protocol extension involving visits every 4 months for five years after initial raltegravir exposure. Participants who did not continue on study-provided raltegravir were followed with annual visits for five years after initial raltegravir exposure (i.e. 48 weeks of raltegravir treatment plus 4 years follow-up). At each visit, a physical exam, blood collection, and determination of treatment adherence occurred. At some visits, urine collection and Tanner staging occurred. Selected cohorts underwent a taste evaluation at 1 of 2 visits. Participants aged 2 to less than 6 years of age were asked to participate in an additional PK substudy in which blood was collected two times over a 12-hour visit (or, if more convenient, this assessment may have been completed in 2 separate visits) in order to collect additional Cmin PK data. Participants were re-registered into the same cohort if a dose change was recommended.

Current pediatric Food and Drug Administration approval and dosing recommendations are based upon evaluations in 122 Final Dose participants aged ≥4 weeks to 18 years enrolled in this study.

The results present safety and efficacy results of the complete 5 year follow up data (primary and key secondary endpoints) of the participants from IMPAACT P1066, the Final Dose Population. By the date on which most of the data were frozen, 24 July 2017, all participants enrolled had Week 24 data (i.e., had either completed the Week 24 visit, or, for those who discontinued before Week 24, had the potential to have experienced the Week 24 visit), had also completed (or had the potential to have experienced) the Week 48 visit, and had either completed 240 weeks of study and were subsequently taken off study, or had prematurely discontinued study and were no longer in follow up.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Documentation of HIV-1 infection, defined as positive results from two samples collected at different time points. More information on this criterion can be found in the protocol.
* For participants in Cohorts I, IIA, IIB, and III: On unchanged therapeutic regimen for at least 12 weeks, or treatment experienced (not including therapy to interrupt maternal-to-child-transmission (MTCT)) but on no treatment for 4 or more weeks prior to study entry. More information on this criterion can be found in the protocol.
* Participants in Cohorts IV must have received therapy to either interrupt MTCT and/or to treat HIV infection and participants in Cohort V must have received therapy to interrupt MTCT but have not received other anti-HIV therapies.
* HIV RNA (ribonucleic acid) of 1,000 copies/mL or greater at screening
* Demonstrated ability or willingness to take assigned raltegravir preparation
* Parent or legal guardian or participant able and willing to provide signed informed consent when applicable
* Female participants who are sexually active and potentially able to become pregnant must use two methods of birth control while on study and for 3 months after stopping study drug. More information on this criterion can be found in the protocol. Male participants must not participate in sperm donation programs. Male participants engaging in sexual activity that could lead to pregnancy must use a condom.
* Willing to be re-registered within same cohort if a dose change is recommended

Exclusion Criteria for All Participants:

* Known Grade 3 or higher of any of the following laboratory tests within 30 days prior to study entry: neutrophil count, hemoglobin, platelets, aspartate aminotransferase (AST), alanine aminotransferase (ALT), lipase, serum creatinine
* Clinical evidence of pancreatitis
* Treatment for active tuberculosis (TB) infection or disease.
* History of lactic acidosis in 3 months prior to study entry. More information on this criterion can be found in the protocol.
* Diagnosis of new Centers for Disease Control Stage C criteria or opportunistic or bacterial infection diagnosed within 30 days prior to study screening and not considered clinically stable
* Prior treatment with another experimental HIV integrase inhibitor
* Immunosuppressive therapy within 30 days prior to beginning raltegravir study treatment. Participants taking short courses of corticosteroids are not excluded.
* Current or anticipated use of any disallowed medications, listed in the protocol.
* Any history of malignancy
* Participants who are unlikely to adhere to the study procedures or keep appointments
* Participants who are planning to relocate during study
* Any clinically significant diseases (other than HIV) or findings during the screening medical history or physical examination that, in the opinion of the investigator, would compromise the outcome of the study
* Current or past participation in an investigational study with a compound or device that is not commercially available within 30 days of signing informed consent
* Participants who are pregnant or breastfeeding. Infants who are receiving breastmilk are allowed to enroll.
* For participants in Cohorts IV and V, participant's caregiver is unable to access clean water supply (as defined by local standards) to re-suspend raltegravir oral granules

Exclusion Criteria for Stage I Participants:

* Stage I mini cohort (initial 4 participants) only: current or anticipated use of antiretroviral regimen that includes atazanavir, tenofovir, or tipranavir during Stage I. Any other commercially available antiretroviral drugs are acceptable.
* Stage I participants enrolling after initial 4 participants: use of atazanavir, tenofovir, or tipranavir prior to the intensive PK testing. More information on this criterion can be found in the protocol.

Exclusion Criteria for Stage II Participants Taking Atazanavir as Part of Their Background Regimen:

* Total bilirubin of Grade 4 or higher within 30 days of study entry
* Total bilirubin value lower than Grade 4 but direct bilirubin or concurrent transaminase greater than 1.5 times the upper limit of normal and participant is symptomatic, within 30 days prior to study entry

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Nachman, MD, Study Chair — State University of New York at Stony Brook, Health Science Center; Andrew Wiznia, MD, Study Chair — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (42):
- United States (29):
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Children's Hospital of Los Angeles NICHD CRS, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Philadelphia IMPAACT Unit CRS, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Hosp. General de Agudos Buenos Aires Argentina NICHD CRS, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Gaborone CRS, Gaborone, Botswana
- Brazil (6):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora da Conceicao NICHD CRS, Porto Alegre, Rio Grande do Sul
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Inst de Infectologia Emilio Ribas Sao Paulo Brazil NICHD CRS, São Paulo
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Shandukani Research CRS, Johannesburg, Gauteng
  - Durban Paediatric HIV CRS, Durban, KwaZulu-Natal
  - Family Clinical Research Unit (FAM-CRU) CRS, Tygerberg, Western Cape

REFERENCES:
- [Background] Cooper D, Gatell J, Rockstroh J, Katlama C, Yeni P, Lazzarin A, Chen J, Isaacs R, Teppler H, Nguyen B, and for the BENCHMRK-1 Study Group. Results of BENCHMRK-1, a Phase III Study Evaluating the Efficacy and Safety of MK-0518, a Novel HIV-1 Integrase Inhibitor, in Patients with Triple-class Resistant Virus. 14th Conference on Retroviruses and Opportunistic Infections, Los Angeles, CA, Abstract 105aLB, 2007.
- [Background] Dayam R, Al-Mawsawi LQ, Neamati N. HIV-1 integrase inhibitors: an emerging clinical reality. Drugs R D. 2007;8(3):155-68. doi: 10.2165/00126839-200708030-00003. PMID 17472411
- [Background] Markowitz M, Morales-Ramirez JO, Nguyen BY, Kovacs CM, Steigbigel RT, Cooper DA, Liporace R, Schwartz R, Isaacs R, Gilde LR, Wenning L, Zhao J, Teppler H. Antiretroviral activity, pharmacokinetics, and tolerability of MK-0518, a novel inhibitor of HIV-1 integrase, dosed as monotherapy for 10 days in treatment-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2006 Dec 15;43(5):509-15. doi: 10.1097/QAI.0b013e31802b4956. PMID 17133211
- [Background] Nair V, Chi G. HIV integrase inhibitors as therapeutic agents in AIDS. Rev Med Virol. 2007 Jul-Aug;17(4):277-95. doi: 10.1002/rmv.539. PMID 17503547
- [Result] Sharon Nachman, Edward Acosta, Nan Zheng, Hedy Tepler, Brenda Homony, Terence Fenton, Edward Handelsman, Carol Worrell, Bobbie Graham, Andrew Wiznia , and the P1066 Group. Interim Results for IMPAACT P1066 Raltegravir (RAL) Oral Chewable Tablet (CT) Formulation on Children 2-5 Years. CROI 2011, Boston, MA, Feb27-March2, 2011.
- [Result] S. Nachman, E. Acosta, N. Zheng, H. Teppler, B. Homony, X. Xu, C. Alvero, E. Handelsman, C. Worrell, B. Graham, M. Toye, A. Wiznia, and the P1066 Group. IMPAACT P1066: Raltegravir (RAL) safety and efficacy in treatment experienced HIV infected (+) youth 2 to 18 years of age through week 48. XIX International AIDS Conference, July 22-27, 2012, Washington, DC.
- [Result] Julie Nelson, A Loftis, K Below, D Cole, S Nachman, L Frenkel, C Alvero, N Zheng, J Eron, and S Fiscus. Absence of Integrase Inhibitor Resistance Mutations in Children Not Treated with Integrase Inhibitor. CROI 2012, Seattle, WA. March 2012.
- [Result] Nachman S, Zheng N, Acosta EP, Teppler H, Homony B, Graham B, Fenton T, Xu X, Wenning L, Spector SA, Frenkel LM, Alvero C, Worrell C, Handelsman E, Wiznia A; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) P1066 Study Team. Pharmacokinetics, safety, and 48-week efficacy of oral raltegravir in HIV-1-infected children aged 2 through 18 years. Clin Infect Dis. 2014 Feb;58(3):413-22. doi: 10.1093/cid/cit696. Epub 2013 Oct 21. PMID 24145879
- [Derived] Nachman S, Alvero C, Teppler H, Homony B, Rodgers AJ, Graham BL, Fenton T, Frenkel LM, Browning RS, Hazra R, Wiznia AA; IMPAACT 1066 study team. Safety and efficacy at 240 weeks of different raltegravir formulations in children with HIV-1: a phase 1/2 open label, non-randomised, multicentre trial. Lancet HIV. 2018 Dec;5(12):e715-e722. doi: 10.1016/S2352-3018(18)30257-1. PMID 30527329
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004; Clarification, August 2009 — https://rsc.tech-res.com/docs/default-source/safety/table_for_grading_severity_of_adult_pediatric_adverse_events.pdf?sfvrsn=6
- See also: Description: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=10

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I: Participants between the ages of 12 and 18 years; receiving raltegravir poloxamer film coated tablet; final selected dose: 400-mg tablet taken orally twice daily.
- Cohort IIA: Participants between the ages of 6 and 11 years; receiving raltegravir poloxamer film coated tablet: final selected dose: 400-mg tablet taken orally twice daily for participants weighing at least 25 kg.
- Cohort IIB: Participants between the ages of 6 and 11 years; receiving raltegravir chewable tablet: final selected dose: Weight based dose of ~6 mg/kg to a maximum dose of 300 mg, taken orally twice daily.
- Cohort III: Participants between the ages of 2 and 5 years; receiving raltegravir chewable tablet: final selected dose: Weight based dose of ~6 mg/kg to a maximum dose of 300 mg, taken orally twice daily.
- Cohort IV: Participants between the ages of 6 and 23 months; receiving raltegravir oral granules for suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data.
- Cohort V: Participants between the ages of 4 weeks and 5 months; receiving raltegravir oral granules for suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data.
Period: Overall Study
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Started | 71 | 16 | 18 | 21 | 15 | 12
Completed Week 24 | 67 | 16 | 18 | 21 | 14 | 11
Completed | 35 | 9 | 12 | 17 | 9 | 5
Not Completed | 36 | 7 | 6 | 4 | 6 | 7
Not completed — Enrolled But Not Given Treatment | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 3 | 1 | 3
Not completed — Pregnancy | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Disallowed Medication | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Number/Volume/Timing of Study Meds | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Guardian Consent Withdrawn | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Intolerance/Unable to Tolerate Dose | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Not Able to Attend Clinic | 5 | 0 | 0 | 1 | 1 | 2
Not completed — Non-Compliant | 17 | 2 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0 | 0 | 1
Not completed — Other Reason | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Population: All patients exposed to raltegravir (at any dose)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V | Total
Number analyzed (Participants) | 71 | 16 | 18 | 21 | 14 | 12 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2) | 9.1 (1.6) | 8.9 (1.6) | 3.1 (1.2) | 1.0 (0.5) | 0.3 (0.1) | 9.5 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 7 | 7 | 13 | 5 | 4 | 70
  Male | 37 | 9 | 11 | 8 | 9 | 8 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 4 | 12 | 8 | 5 | 0 | 55
  Not Hispanic or Latino | 43 | 11 | 6 | 10 | 3 | 8 | 81
  Unknown or Not Reported | 2 | 1 | 0 | 3 | 6 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 42 | 12 | 7 | 14 | 10 | 12 | 97
  White | 25 | 3 | 10 | 5 | 2 | 0 | 45
  More than one race | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 3 | 1 | 1 | 1 | 1 | 0 | 7
Plasma HIV RNA, continuous [Mean (Standard Deviation); unit: log10 copies/mL] | 4.3 (0.6) | 4.3 (0.6) | 4.3 (0.5) | 4.4 (0.8) | 5.4 (1) | 6 (1.2) | 4.6 (0.9)
Plasma HIV RNA, categorical [Number; unit: participants]
  0 to ≤4,000 copies/mL | 10 | 2 | 2 | 2 | 1 | 0 | 16
  >4,000 to ≤50,000 copies/mL | 40 | 12 | 11 | 11 | 1 | 2 | 74
  >50,000 to ≤100,000 copies/mL | 14 | 1 | 4 | 4 | 3 | 1 | 23
  >100,000 copies/mL | 7 | 1 | 1 | 4 | 9 | 9 | 13
CD4 cell count [Mean (Standard Deviation); unit: cells/µL] | 410.7 (238.2) | 652.3 (360.4) | 545.4 (280.2) | 1122.9 (537.1) | 1647.5 (965.7) | 1359.6 (1003.8) | 744.3 (654.9)
CD4 percentage [Mean (Standard Deviation); unit: Percentage of total lymphocytes] | 19.9 (9.6) | 25.4 (8.2) | 26.7 (10.6) | 27.9 (8.2) | 22.6 (8.1) | 18.4 (11.5) | 23 (9.9)
CDC HIV Clinical Classification [Number; unit: participants] — The CDC Classification System for HIV Infection is the medical classification system used by the United States Centers for Disease Control and Prevention (CDC) to classify HIV disease and infection. http://www.cdc.gov/mmwr/preview/mmwrhtml/00032890.htm
  participants
    A | 17 | 5 | 6 | 5 | 6 | 4 | 33
    B | 29 | 3 | 5 | 1 | 2 | 1 | 38
    C | 24 | 7 | 2 | 8 | 3 | 0 | 41
    N | 1 | 1 | 5 | 7 | 3 | 7 | 14
Number of antiretroviral (ARV) classes previously used [Number; unit: participants]
  0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  1 | 2 | 0 | 0 | 2 | 8 | 10 | 4
  2 | 9 | 5 | 8 | 13 | 4 | 2 | 35
  ≥3 | 60 | 11 | 10 | 5 | 2 | 0 | 86
Duration of ARVs previously used [Mean (Standard Deviation); unit: years] | 12 (3.8) | 8.5 (2.3) | 7.1 (3) | 2.4 (1.4) | 0.4 (0.5) | 0.1 (0.1) | 7.7 (5.6)
Prior use of Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI) [Number; unit: participants]
  Yes | 60 | 14 | 15 | 10 | 8 | 11 | 118
  No | 11 | 2 | 3 | 11 | 6 | 1 | 34
Use of prior PIs [Number; unit: participants]
  Yes | 69 | 13 | 13 | 13 | 5 | 0 | 113
  No | 2 | 3 | 5 | 8 | 9 | 12 | 39
Phenotypic Sensitivity score [Number; unit: participants] — The Phenotypic Sensitivity score (PSS) was defined as the total number of ARVs in optimized background therapy (OBT) to which the subject's viral isolate showed phenotypic sensitivity, based on pre-study resistance tests. The PSS score range is from 0 (meaning there was no ARV the subject was sensitive to) to >=3 (the subject was sensitive to >=3 of the ARVs in his/her OBT). If no resistance results were available for a drug, it was scored as one active drug in the PSS if there was history of prior use, and was considered not active if no prior use. Scoring did not include Raltegravir.
  participants
    0 | 5 | 1 | 0 | 0 | 0 | 0 | 6
    1 | 15 | 4 | 7 | 2 | 0 | 1 | 29
    2 | 25 | 2 | 8 | 8 | 2 | 5 | 50
    ≥3 | 21 | 7 | 2 | 6 | 9 | 4 | 49
    Missing | 5 | 2 | 1 | 5 | 3 | 2 | 18
Genotypic sensitivity score [Number; unit: participants] — The Genotypic Sensitivity score (GSS) was defined as the total number of ARVs in OBT to which the subject's viral isolate showed genotypic sensitivity, based on pre-study resistance tests. The GSS score range is from 0 (meaning there was no ARV the subject was sensitive to) to >=3 (the subject was sensitive to >=3 of the ARVs in his/her OBT). If no resistance results were available for a drug, it was scored as one active drug in the GSS if there was history of prior use, and was considered not active if no prior use. Scoring did not include Raltegravir.
  participants
    0 | 9 | 1 | 0 | 0 | 0 | 0 | 10
    1 | 23 | 4 | 9 | 2 | 0 | 1 | 39
    2 | 20 | 6 | 7 | 11 | 3 | 5 | 52
    ≥3 | 18 | 5 | 2 | 7 | 10 | 3 | 45
    Missing | 1 | 0 | 0 | 1 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or 4 Adverse Events (AEs)
Description: Adverse events were graded using the Division of AIDS (DAIDS) AE Grading Table, Version 1.0. All grade 3 and higher signs, symptoms, and laboratory toxicities were included.
Time Frame: From study entry through Week 24
Population: Final Dose Population: Participants accrued into Stage I and treated only at the dose ultimately selected for their cohorts were combined with those accrued into Stage II, where all participants received only the final selected doses for their respective cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
percentage of participants | 20.3 [11 to 32.8] | 25 [0.6 to 80.6] | 15.4 [1.9 to 45.4] | 30 [11.9 to 54.3] | 35.7 [12.8 to 64.9] | 33.3 [9.9 to 65.1]

2. Primary Outcome: Number of Participants Terminated From Treatment Due to Suspected Adverse Drug Reaction (SADR) Attributable to the Study Medication
Description: The attribution of relationship of serious adverse events to study drug for the purposes of employing the start, stop and pause rules was by consensus among the site investigator, study team (which includes representatives from Merck) and the Division of AIDS medical officer; if unanimous agreement between them cannot be established, the attribution made by the majority of these 3 persons or entities will be used. Gradation of relationship will use the following terminology: Not related, Probably not related, Possibly related, Probably related or Definitely related.
Time Frame: From study entry through Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cohort IV: Participants between the ages of 6 and 23 months; receiving raltegravir granules for oral suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died were summarized.
Time Frame: From study entry through Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cohort V: Participants between the ages of 4 weeks and 5 months; receiving raltegravir oral granules for suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data. .
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Curve (AUC12h)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (WinNonlin version 4.01, Pharsight Corp., Mountain View, CA). AUC12h (area-under-the-curve from 0 to 12 hours) were determined using the linear-log trapezoidal rule.
Time Frame: Measured between days 5 and 12 of raltegravir initiation; Blood samples were drawn pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post dosing.
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose (Stage I).
Measure: Mean (Standard Deviation); unit: hour*mg/L
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 8 | 11
hour*mg/L | 10.2 (10.0) | 13.4 (16.1) | 10.5 (3.5) | 9.5 (5.5) | 9.3 (3.2) | 10.9 (4.4)

5. Primary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (WinNonlin version 4.01, Pharsight Corp., Mountain View, CA). Maximum plasma concentration (Cmax) was taken directly from the observed concentration-time data.
Time Frame: as for outcome 4
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose (Stage I).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 8 | 11
ng/mL | 2813.1 (2673.9) | 4055.7 (5269.5) | 5314.2 (2842.6) | 5204.8 (2940.6) | 5683.0 (3685.0) | 4299.0 (1661.9)

6. Primary Outcome: PK Parameter: Time to Half of Maximum Plasma Concentration Cmax (T1/2)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (WinNonlin version 4.01, Pharsight Corp., Mountain View, CA). Time to half of maximum plasma concentration Cmax (T1/2) was taken directly from the observed concentration-time data.
Time Frame: as for outcome 4
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose (Stage I).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 8 | 11
hour | 4.9 (3.6) | 3.7 (1.4) | 4.5 (4.2) | 4.1 (3.2) | 3.0 (1.8) | 2.1 (1.5)

7. Primary Outcome: PK Parameter: Concentration at 12 Hours Postdose (C12h)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using noncompartmental methods (WinNonlin version 4.01, Pharsight Corp., Mountain View, CA). Plasma concentration at 12 hours postdose (C12h) was taken directly from the observed concentration-time data.
Time Frame: as for outcome 4
Population: Participants with intensive pharmacokinetic (PK) results at the final recommended dose (Stage I).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 8 | 11
ng/mL | 197.0 (154.2) | 399.4 (880.9) | 78.7 (68.9) | 39.5 (21.9) | 56.4 (26.8) | 99.6 (83.9)

8. Secondary Outcome: Percentage of Participants With Grade 3 or 4 Adverse Events (AEs)
Description: as for outcome 1
Time Frame: From study entry through Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
percentage of participants | 23.7 [13.6 to 36.6] | 25 [0.6 to 80.6] | 23.1 [5 to 53.8] | 40 [19.1 to 63.9] | 42.9 [17.7 to 71.1] | 33.3 [9.9 to 65.1]

9. Secondary Outcome: Number of Participants Terminated From Treatment Due to Suspected Adverse Drug Reaction (SADR) Attributable to the Study Medication
Description: as for outcome 2
Time Frame: From study entry through Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cohort IV -Data Not Included in This Interim Analysis.: Participants between the ages of 6 and 23 months; receiving raltegravir oral granules for suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data.
- Cohort V -Data Not Included in This Interim Analysis.: Participants between the ages of 4 weeks and 5 months; receiving raltegravir oral granules for suspension (20 mg/mL): Stage I starting dose of 6 mg/kg orally twice daily according to dosing table in protocol or the dose determined by review of all available data.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV -Data Not Included in This Interim Analysis. | Cohort V -Data Not Included in This Interim Analysis.
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died were summarized.
Time Frame: From study entry through Week 48
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With ≥1 log10 Drop From Baseline in HIV RNA or HIV RNA <400 Copies/mL
Description: Plasma HIV RNA concentrations were determined at entry and at regular intervals using the HIV-1 MONITOR Test, version 1.5 (Roche Molecular Diagnostics) or RealTime HIV-1 (Abbott Molecular), and analyses used the Observed Failure Approach.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
percentage of participants
  Baseline to Week 24 | 72.4 [59.1 to 83.3] | 50 [6.8 to 93.2] | 76.9 [46.2 to 95] | 70 [45.7 to 88.1] | 85.7 [57.2 to 98.2] | 100 [71.5 to 100]
  Baseline to Week 48 | 75 [61.6 to 85.6] | 75 [19.4 to 99.4] | 90.9 [58.7 to 99.8] | 84.2 [60.4 to 96.6] | 92.9 [66.1 to 99.8] | 80 [44.4 to 97.5]

12. Secondary Outcome: Change of CD4 Count From Baseline
Description: Change in CD4 cell count from baseline was calculated as the value at later visit minus the value at baseline.
Time Frame: Baseline, Week 24, 48
Population: Final Dose Population: Participants accrued into Stage I and treated only at the dose ultimately selected for their cohorts are combined with those accrued into Stage II, where all participants received only the final selected doses for their respective cohorts.
Measure: Mean (95% Confidence Interval); unit: cells/µL
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
cells/µL
  Baseline to Week 24 | 114.6 [73.9 to 155.4] | -35.8 [-348.8 to 277.3] | 143.4 [-12.9 to 299.6] | 147.2 [-2.7 to 297.1] | 400.5 [60.3 to 740.6] | 499.2 [-50.4 to 1048.7]
  Baseline to Week 48 | 168.4 [117.7 to 219.1] | 189.5 [-154.2 to 533.2] | 76.8 [-85.3 to 238.9] | 158.1 [11.7 to 304.4] | 278.8 [-185.6 to 743.2] | 876.0 [362.7 to 1389.3]

13. Secondary Outcome: Change of CD4 Percent From Baseline
Description: Change in CD4 percent from baseline was calculated as the value of the later visit minus the value at baseline.
Time Frame: Baseline, Week 24, 48
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: percentage of total lymphocytes
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 59 | 4 | 13 | 20 | 14 | 12
percentage of total lymphocytes
  Baseline to Week 24 | 4.1 [2.8 to 5.3] | 2.2 [-7.2 to 11.5] | 0.8 [-3.6 to 5.2] | 5.3 [2.9 to 7.7] | 6.2 [1.3 to 11.2] | 9.0 [4.6 to 13.4]
  Baseline to Week 48 | 5.2 [3.9 to 6.6] | 6.0 [-2.6 to 14.6] | 1.6 [-2.7 to 5.9] | 4.3 [1 to 7.6] | 6.4 [1.4 to 11.3] | 8.7 [2.7 to 14.8]

ADVERSE EVENTS:
Time Frame: From study entry to completion of the study at Week 240 or at 14 days after the premature study discontinuation.
Description: Adverse event summary pertains to the Final Dose Population: participants accrued into Stage I and treated only at the dose ultimately selected for their cohorts werecombined with those accrued into Stage II, where all participants received only the final selected doses for their respective cohorts. The study protocol required reporting of all new diagnoses, signs/symptoms, and laboratory events of >=Grade 1; the protocol team assessed attribution to treatment for adverse events >=Grade 3.
Arm/Group | Cohort I | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/4 | 0/13 | 0/20 | 1/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 26/59 | 2/4 | 4/13 | 7/20 | 7/14 | 4/12
Other Adverse Events (participants affected / at risk) | 57/59 | 4/4 | 13/13 | 20/20 | 14/14 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=59) | Cohort IIA (N=4) | Cohort IIB (N=13) | Cohort III (N=20) | Cohort IV (N=14) | Cohort V (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 0 | 0 | 2 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Lipase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 6 | 0 | 0 | 2 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Treatment noncompliance (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I (N=59) | Cohort IIA (N=4) | Cohort IIB (N=13) | Cohort III (N=20) | Cohort IV (N=14) | Cohort V (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1 | 4 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 9 | 0 | 1 | 7 | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 4 | 0 | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ear canal erythema (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 14 | 0 | 4 | 3 | 2 | 0
Ear pruritus (Ear and labyrinth disorders) | 2 | 0 | 0 | 1 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0
Noninfective myringitis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 4 | 0 | 1 | 3 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 2 | 0 | 1 | 0 | 1 | 0
Tympanosclerosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival pallor (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0
Eye discharge (Eye disorders) | 4 | 0 | 0 | 3 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 5 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 3 | 1 | 1 | 2 | 1 | 2
Eye swelling (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eyelid thickening (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 8 | 0 | 2 | 2 | 1 | 1
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 1 | 1 | 2 | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 8 | 0 | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 1 | 3 | 7 | 9 | 7
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 0 | 2 | 1 | 1 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral discharge (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 1 | 2
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 21 | 0 | 4 | 9 | 6 | 3
Adverse event (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 7 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 3 | 0 | 0 | 0 | 0 | 0
Crepitations (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Crying (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 0 | 2 | 2 | 0 | 0
Influenza like illness (General disorders) | 5 | 0 | 1 | 0 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 5 | 0 | 0 | 1 | 0 | 0
Mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 4 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 2 | 1 | 1 | 0 | 0 | 0
Puncture site discharge (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 28 | 3 | 8 | 9 | 8 | 6
Secretion discharge (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 3 | 2 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 4 | 0 | 1 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 3
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 4 | 1 | 0 | 1 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 4 | 0 | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cervicitis human papilloma virus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cervicitis trichomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chlamydial cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 0 | 2 | 4 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 3 | 6 | 6 | 3
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
HIV associated nephropathy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
HIV wasting syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 5 | 0 | 0 | 1 | 0 | 0
Hymenolepiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 9 | 1 | 1
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 6 | 0 | 0 | 2 | 2 | 1
Oral hairy leukoplakia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 2 | 3 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 8 | 0 | 3 | 9 | 4 | 2
Otitis media acute (Infections and infestations) | 3 | 0 | 1 | 1 | 1 | 0
Otitis media chronic (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Pancreatitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Persistent generalised lymphadenopathy (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Pharyngeal chlamydia infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 0 | 2 | 2 | 6 | 4
Pharyngitis streptococcal (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 4 | 0 | 0 | 0 | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Proctitis chlamydial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Proctitis gonococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Purulent discharge (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Rubella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 2 | 2 | 3 | 5 | 2 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 1 | 0 | 0 | 4 | 2 | 2
Tinea faciei (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Tinea infection (Infections and infestations) | 2 | 0 | 0 | 2 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Urethritis chlamydial (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Urethritis gonococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vaginitis chlamydial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Virologic failure (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis gonococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 0
Genital injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 5 | 0 | 2 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Stoma site rash (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 19 | 1 | 4 | 3 | 5 | 4
Aspartate aminotransferase increased (Investigations) | 15 | 2 | 4 | 4 | 8 | 4
Blood albumin decreased (Investigations) | 12 | 0 | 0 | 3 | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 11 | 1 | 1 | 3 | 0 | 1
Blood bicarbonate decreased (Investigations) | 24 | 0 | 4 | 11 | 8 | 5
Blood bilirubin increased (Investigations) | 13 | 1 | 4 | 0 | 2 | 1
Blood calcium decreased (Investigations) | 4 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 9 | 0 | 3 | 9 | 1 | 0
Blood creatinine increased (Investigations) | 7 | 0 | 1 | 1 | 2 | 0
Blood glucose decreased (Investigations) | 22 | 1 | 7 | 8 | 5 | 1
Blood glucose increased (Investigations) | 14 | 1 | 1 | 3 | 9 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pH increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 14 | 2 | 3 | 1 | 4 | 2
Blood potassium decreased (Investigations) | 15 | 2 | 1 | 2 | 5 | 2
Blood potassium increased (Investigations) | 0 | 1 | 0 | 4 | 7 | 9
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood sodium abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 28 | 2 | 6 | 14 | 9 | 10
Blood sodium increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 3 | 0 | 2 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 8 | 0 | 1 | 2 | 6 | 9
Helicobacter test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 9 | 0 | 1 | 2 | 2 | 3
Low density lipoprotein increased (Investigations) | 8 | 0 | 1 | 8 | 0 | 0
Neutrophil count decreased (Investigations) | 18 | 1 | 5 | 8 | 11 | 2
Platelet count decreased (Investigations) | 7 | 0 | 3 | 1 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Viral load increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 0 | 0 | 1 | 3 | 1
White blood cell count decreased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Body fat disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 3 | 3 | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 3
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Head deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2 | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dyscalculia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyslalia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 25 | 4 | 2 | 1 | 1 | 0
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0
Language disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Meningeal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
First trimester pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 6 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Learning disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Oppositional defiant disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Reading disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sexually inappropriate behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep terror (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 0
Kidney enlargement (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 4 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Male sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Perineal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 6 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 2 | 0
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 2 | 6 | 15 | 9 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 2 | 1 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 29 | 2 | 7 | 7 | 6 | 9
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nasal turbinate abnormality (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 0 | 5 | 2 | 1 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1 | 1 | 0
Pharyngeal exudate (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25 | 1 | 6 | 12 | 6 | 10
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 2 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 | 1 | 3 | 4 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 9 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 3 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 2 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 7 | 1 | 1 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 3 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 0 | 2 | 2 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 1 | 5 | 7 | 9
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 2 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 6 | 0 | 0 | 3 | 1 | 2
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0
Victim of sexual abuse (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights